CLINICAL TRIAL: NCT02150122
Title: A Dose-response, Double-blind Randomised Placebo-controlled Trial to Estimate the Dietary Requirement for Vitamin D in Caucasian Male and Female Adolescents Aged 14-18 Years (The ODIN Study)
Brief Title: Dietary Requirement for Vitamin D in Adolescents Aged 14-18 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ODIN/1213
Record Dates: First submitted 2014-05-23; First posted 2014-05-29 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Serum 25-hydroxyvitamin D Concentrations (25OHD)
Keywords: Vitamin D; Serum 25-hydroxyvitamin D (25OHD); Adolescents
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 10 micrograms (400 IU) vitamin D3 (Experimental): Participants will be given a daily supplement containing 10 micrograms (400 IU) vitamin D3 to take for 5 months.
  Interventions: Dietary Supplement: Vitamin D3
- 20 micrograms (800 IU) vitamin D3 (Experimental): Participants will be given a daily supplement containing 20 micrograms (800 IU) vitamin D3 to take for 5 months.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (No Intervention): Participants will be given a placebo, similar in appearance to the vitamin D3 tablets, to take for 5 months.

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Arms: 10 micrograms (400 IU) vitamin D3; 20 micrograms (800 IU) vitamin D3

SUMMARY:
It is known that low vitamin D status is a very common problem in the UK. It is also known that a lack of vitamin D availability has potentially serious health implications, especially with respect to bone and muscle function. Much research has recently taken place to establish the vitamin D requirements of key population groups (i.e. pregnant women, the elderly, ethnic minorities). However few data are available describing the vitamin D requirements for male and female adolescents. The period of adolescence is a key stage of growth and development - poor nutrition during this time can have detrimental health consequences for a lifetime.

No intervention studies have comprehensively investigated the vitamin D requirements of adolescents. The proposed ODIN Study will enable a better understanding of how adolescents respond to vitamin D supplementation and the most effective daily amount that will raise and maintain vitamin D status in adolescents during the winter-time. In addition, investigations into the mechanisms of action with respect to any differences observed across the doses of vitamin D and between the genders of the participants will also provide key information. Mechanisms of action will focus on genetic differences as well as differences in vitamin D metabolising enzymes.

The results obtained from this significant study will not only inform the European Food Standards Agency (EFSA) with respect to their imminent deliberations regarding vitamin D recommendations. The ODIN Study will also inform the UK Department of Health's Scientific Advisory Committee on Nutrition (SACN), the wider scientific community and be a critical resource for key stakeholders (i.e. food industry, government health agencies) to collaborate in determining future public health strategies, thus potentially positively impacting on the health of the population for years to come.

The investigators propose that the daily supplementation of 10µg/day (400 IU) and 20µg/day (800 IU) of vitamin D3 for five months will meet the vitamin D requirements of males and females aged 14-18 year and will be sufficient to maintain winter-time 25OHD levels above a range of thresholds between 30 and 50nmol/l.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged between 14 and 18 years
* Caucasian ethnicity
* In good health
* Written informed consent from the adolescent (and parent if required)

Exclusion Criteria:

* Currently receiving treatment for medical conditions likely to affect vitamin D metabolism
* Hypercalcaemia (>2.5mmol/l)
* Regular use of sun-beds
* Having a sun holiday one month prior to commencing the trial or plans for a sun holiday within the study period.
* Use of vitamin supplements containing vitamin D - if the prospective participant agrees to stop vitamin D supplementation to join the study, a wash-out period of 8 weeks prior to commencing the trial would be acceptable.
* Excessive consumption of alcohol (>14 units per week for females, >21 units per week for males)
* Smoking >10 cigarettes per day
* Those following a weight-reducing diet or under dietary restriction (except vegetarianism)
* Known intolerance/allergy to the constituent ingredients of the daily supplement
* Clinically significant haematological abnormalities other than mild anaemia (Hb<12.0g/dl)
* Active malignancy
* Pregnant or planning a pregnancy during the study period.
* Breast-feeding mothers

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D concentrations | Baseline and after 5 months of supplementation
  To investigate the vitamin D intakes needed to maintain serum 25-hydroxyvitamin D (25OHD) concentrations above the deficiency and insufficiency cut off thresholds (30nmol/l and 50nmol/l respectively) in male and female adolescents during the winter time.

OTHER OUTCOMES:
Identification of genetic polymorphisms for vitamin D | Baseline and after 5 months of supplementation
  To investigate the mechanisms (genetic/enzymatic) underlying the differences observed in the preceding objective via genotyping the participants for polymorphisms related to vitamin D metabolism. Secondary analyses will include evaluation of variations in the response to supplementation by single SNP variations and by the genetic vitamin D risk score. To determine, through transcriptomic (global mRNA) analysis of leukocyte samples, genome-wide differences in gene expression, in the adolescents in response to the vitamin D3 supplementation.
Family links in vitamin D levels and bone health | Baseline
  To determine the bone mineral density and vitamin D levels (in addition to the assessment of related blood markers and lifestyle factors) of the mothers of the adolescent participants, in order to establish possible familial links in the factors that affect vitamin D status and bone health.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Lanham-New, Professor, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Smith TJ, Tripkovic L, Hauger H, Damsgaard CT, Molgaard C, Lanham-New SA, Hart KH. Winter Cholecalciferol Supplementation at 51 degrees N Has No Effect on Markers of Cardiometabolic Risk in Healthy Adolescents Aged 14-18 Years. J Nutr. 2018 Aug 1;148(8):1269-1275. doi: 10.1093/jn/nxy079. PMID 29920594
- [Derived] Smith TJ, Tripkovic L, Damsgaard CT, Molgaard C, Ritz C, Wilson-Barnes SL, Dowling KG, Hennessy A, Cashman KD, Kiely M, Lanham-New SA, Hart KH. Estimation of the dietary requirement for vitamin D in adolescents aged 14-18 y: a dose-response, double-blind, randomized placebo-controlled trial. Am J Clin Nutr. 2016 Nov;104(5):1301-1309. doi: 10.3945/ajcn.116.138065. Epub 2016 Sep 21. PMID 27655438